CLINICAL TRIAL: NCT06269341
Title: Long-term Outcomes of Smoker and Drinker With Esophageal Squamous Cell Carcinoma After Esophagectomy
Brief Title: Outcomes of Smoker and Drinker With Esophageal Squamous Cell Carcinoma After Esophagectomy
Acronym: OSinEC
Status: Recruiting | Type: Observational
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yongtao Han, MD, Sichuan Cancer Hospital and Research Institute
Other Study IDs: SCCH-TS2208
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Outcomes of Smoker and Drinker After Esophagectomy
Keywords: survival; esophgeal cancer; smoker; drinker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high-risk: Smoker and Drinker with Esophageal Squamous Cell Carcinoma after Esophagectomy
  Interventions: Other: No intervention
- low-risk: Non-Smoker and Non-Drinker with Esophageal Squamous Cell Carcinoma after Esophagectomy

INTERVENTIONS:
Other: No intervention — No intervention
  Groups: high-risk

SUMMARY:
Our study demonstrates that patients who did not consume alcohol or smoke had a significant advantage in overall survival (OS) after undergoing esophagectomy. Furthermore, our findings indicate that there was no statistically significant difference in OS between patients with a history of both smoking and drinking, and those who only smoked or drank

ELIGIBILITY:
Inclusion Criteria:

patients with esophageal cancer

Exclusion Criteria:

(1) pathology confirmed a non-squamous cell carcinoma, (2) the tumor was located outside of the thoracic region, (3) R1/R2 resection was performed indicating incomplete tumor removal, (4) evidence of distant tumor metastasis was observed, (5) they underwent preoperative neoadjuvant therapy, (6) pTis/T1a stage (7) Missing data.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with esophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 2957 (Estimated)
Dates: Start 2010-02-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | April 2022-April 2024
  Overall Survival was calculated from the month and year of surgery to the time of death or last follow-up in April 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No